CLINICAL TRIAL: NCT00748852
Title: An Eight Week, Open-label Extension Study Evaluating the Safety of JTT-302 Administered Once Daily in Subjects With Low HDL-C Levels Who Have Completed the Treatment Phase of Study AT302-U-06-003
Brief Title: Safety Study of JTT-302 in Subjects With Low HDL-C Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT302-U-06-004
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): JTT-302, 400 mg
  Interventions: Drug: JTT-302

INTERVENTIONS:
Drug: JTT-302 — JTT-302, 100 mg tablets, 400 mg dose, oral, 30 minutes after the start of the morning meal

SUMMARY:
The purpose of this study is to evaluate the safety of JTT-302 when administered for eight or 12 weeks in subjects with low HDL-C levels and to determine the effect of JTT-302 on lipid parameters and CETP activity and mass.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have successfully completed the 4-week treatment period of study AT302-U-06-003

Exclusion Criteria:

* Females who are pregnant or lactating, and females of child bearing potential who are not using an effective method of contraception
* Use of Cytochrome P450 3A4 inducers or inhibitors, as defined in the protocol
* Subjects who cannot follow the prescription and OTC medication restrictions defined in the protocol
* Flu-shots not permitted during the study, including the follow-up period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety profile of JTT-302 when administered for 8 weeks or 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Percent change and change from baseline after four, eight or 12 weeks exposure to JTT-302 in Lipid Parameters | 4, 8 or 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Ana, California, United States